CLINICAL TRIAL: NCT03964142
Title: Randomized Controlled Trial on Comprehensive Exercise-based Cardiac Rehabilitation Programs for the Prevention of Anthracyclines and/or Anti-HER2 Antibodies-induced Cardiotoxicity in Breast Cancer
Brief Title: Exercise-based Cardiac Rehabilitation for the Prevention of Breast Cancer Chemotherapy-induced Cardiotoxicity
Acronym: ONCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Carlos Peña Gil, Head of the Cardiac Rehabilitation Unit, Cardiology Department, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI17/01687
Record Dates: First submitted 2019-02-21; First posted 2019-05-28 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Cardiotoxicity; Cardiac Rehabilitation
Keywords: Chemotherapy; Anthracyclines; Trastuzumab; Pertuzumab; Antibodies, Monoclonal, Humanized; Breast Cancer; Exercise therapy
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation (Experimental): Patients enrolled in the integrated exercise-based cardiac rehabilitation program (centre-based or telematic)
  Interventions: Other: Cardiac rehabilitation
- Conventional management (No Intervention): Patients with conventional management and physical activity recommendation

INTERVENTIONS:
Other: Cardiac rehabilitation — Integrated cardiac rehabilitation program that includes supervised exercise training*.
  * Due to the COVID-19 pandemic, supervised physical exercise training had to be conducted telematically (through live guided training sessions conducted online, with the same design, frequency, and dosage of exercise).
  Arms: Cardiac Rehabilitation

SUMMARY:
This project aims to determine whether a comprehensive cardiac rehabilitation program including supervised exercise training is able to prevent cardiotoxicity during treatment with anthracyclines and / or anti-HER-2 antibodies in women with breast cancer. Participants will be randomly allocated to cardiac rehabilitation (intervention group) or conventional management with physical exercise recommendation (control group).

DETAILED DESCRIPTION:
Cardiovascular toxicity caused by chemotherapy is the leading cause of death in patients who survive cancer. Physical exercise during chemotherapy has shown to improve quality of life and decrease the risk of death. The objective of this project is to determine whether an intervention through a comprehensive cardiac rehabilitation program including supervised physical exercise is able to prevent anthracyclines and / or anti-HER-2 antibodies-induced cardiotoxicity in women with breast cancer.

For this purpose, the investigators intend to conduct a randomized controlled study including female patients managed under the same cardiotoxicity prevention protocol (clinical, laboratory and echocardiographic follow-up assessment). Patients will be randomized to a non-pharmacological intervention (participation in a multidisciplinary cardiac rehabilitation program with supervised exercise training) or control (conventional management and physical activity recommendation)*.

The investigators hypothesize that a cardiac rehabilitation program may limit chemotherapy-induced cardiotoxicity in women with breast cancer, improve cardiac remodeling assessed by echocardiography and enhance their global cardiovascular risk profile to a greater extent, compared to control group.

* OF NOTE: Due to the COVID-19 pandemics, several modifications to the original protocol were introduced for safety reasons or motivated by the health situation, namely:

1. Intervention: Change from centre-based to telematic supervised exercise training sessions provided within the cardiac rehabilitation program (intervention group)
2. Secondary outcome 4: Change in functional capacity assessed by conventional ergometry or cardiopulmonary exercise test OR the 6-minute walking test (metabolic equivalents: METs or peak oxygen consumption: VO2)
3. Recruiting centres: One centre (Hospital Universitari Vall d'Hebron) withdrew from the study due to the impossibility of assuming its execution.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of breast cancer at early stages (I, II, III)
* Treatment with anthracyclines and / or anti-HER-2 antibodies (trastuzumab and / or pertuzumab)
* Possibility of completing a cardiac rehabilitation program (centre-based or telematic) and programmed visits.
* Providing written informed consent.

Exclusion Criteria:

* Patients with previous history of heart disease or heart failure.
* Left ventricular dysfunction (left ventricular ejection fraction <53%) at baseline.
* Metastatic disease.
* Patients carrying an implantable cardioverter defibrillator.
* Patients with physical or mental limitation to carry out an exercise program.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 122 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular systolic function quantified by left ventricular ejection fraction and global longitudinal strain by transthoracic echocardiography | Baseline to every 3 months through study completion, at the end of the study at an average of 18 months, and every year after study completion up to a maximum of 5 years
  Fall of 10 absolute percentage points of left ventricular ejection fraction with final value below 53% or global longitudinal strain fall >15% with respect to baseline

SECONDARY OUTCOMES:
Change in health-related quality of life assessed by the Functional Assessment of Cancer Therapy - Breast plus Arm Morbidity (FACT-B+4) questionnaire | Baseline and at the end of the study at an average of 18 months
  Score achieved in the Functional Assessment of Cancer Therapy - Breast plus Arm Morbidity (FACT-B+4) questionnaire, a specific validated scale to assess quality of life of women with breast cancer. It comprises 27 items within 5 areas of assessment: physical well-being (7 items), social and family environment (7 items), emotional well-being (7 items), functional well-being (6 items) and worries related to the diagnosis and treatment of the disease (9 items). Each item is scored by means of a Likert scale from 0 to 5, with higher scores representing better results. The total score is obtained by adding the scores for each item, and ranges from a minimum of 0 (worst posible result) to a maximum of 146 (best possible result).
Change in tolerance to chemotherapy: number of participants with significant cardiovascular and non-cardiovascular adverse effects throughout the study | Every 3 months during study completion and at the end of the study at an average of 18 months
  Significant cardiovascular and non-cardiovascular adverse effects during treatment, threatening life, requiring admission, prolonging hospitalization, being clinically relevant or causing chemotherapy interruptions
Change in global functional capacity assessed by conventional ergometry, cardiopulmonary exercise testing (CPET) or the 6-minute walking test (6MWT). | Baseline and at the end of the study at an average of 18 months
  Change in functional capacity assessed by conventional ergometry, cardiopulmonary exercise test or the 6-minute walking test (6MWT) (metabolic equivalents: METs or peak oxygen consumption: VO2) * .
  *Due to COVID-19 pandemic, participants' assessment with CPET had to be stopped for safety concerns. In such cases, functional capacity was estimated from the maximum work rate in the 6-minute walking test (6MWT). This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes, which is well correlated with VO2. The 6MWT has been proved to be valid and reliable for functional capacity assessment in the study population.
Change in localized lower limb functional capacity assessed by number of repetitions performed within 30 seconds in the sit-to-stand test | Baseline and at the end of the study at an average of 18 months
  Number of repetitions in the sit-to-stand test within 30 seconds
Change in shoulder functional capacity assessed by range of degrees in shoulder movement by goniometry | Baseline and at the end of the study at an average of 18 months
  Range of degrees in shoulder movement measured by goniometry
Change in upper limb strength measured by dynamometry (kg) | Baseline and at the end of the study at an average of 18 months
  Kilograms by dynamometry of right and left upper limbs
Change in shoulder pain and disability assessed by the SPADI (shoulder pain and disability index (SPADI) questionnaire | Baseline and at the end of the study at an average of 18 months
  Score achieved in the SPADI (shoulder pain and disability index) questionnaire. The pain dimension consists of five questions regarding the severity of an individual's pain, functional activities are assessed with eight questions. Each question may be scored from 0 to 10. Verbal anchors for the pain dimension are 'no pain at all' (0) and 'worst pain imaginable' (10) ,and those for the functional activities are 'no difficulty' (0) and 'so difficult it required help' (10). The scores from both dimensions are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Change in cardiovascular risk profile as assessed by the presence or absence of classic cardiovascular risk factors | Baseline and at the end of the study at an average of 18 months
  Dyslipidemia, Diabetes mellitus, Arterial Hypertension, Smoking status
Change in anthropometric parameters: height in cm | Baseline and at the end of the study at an average of 18 months
  Height measured in cm
Change in anthropometric parameters: weight in kg | Baseline and at the end of the study at an average of 18 months
  Weight measured in kg
Change in anthropometric parameters: body mass index (BMI) in kg/m^2 | Baseline and at the end of the study at an average of 18 months
  Weight and height will be combined to report BMI in kg/m^2
Change in anthropometric parameters: abdominal circumference in cm | Baseline and at the end of the study at an average of 18 months
  Abdominal perimeter measured with a tape measure in cm
Change in resting heart rate measured by pulse oximetry (beats per min) | Baseline and at the end of the study at an average of 18 months
  Resting heart rate by pulse oximetry (beats per min)
Change in resting blood pressure (mmHg) measured by sphygmomanometer | Baseline and at the end of the study at an average of 18 months
  Resting blood pressure by sphyngomanometer in mmHg
Change in biomarkers NT-ProBNP | Baseline and at the end of the study at an average of 18 months
  Value of NT-ProBNP(pg/mL) in blood tests
Change in biomarkers: troponin | Baseline and at the end of the study at an average of 18 months
  Value of troponin I (ng/mL) in blood tests
Change in biomarkers: haemoglobin | Baseline and at the end of the study at an average of 18 months
  Value of haemoglobin (g/dL) in blood tests
Change in dietary pattern as assessed by the PREDIMED (PREvención con DIeta MEDiterránea) questionnaire | Baseline and at the end of the study at an average of 18 months
  Validated questionnaire to assess adherence to Mediterranean diet, including 14 questions regarding dietary habits, rated with 0 or +1 points. Global score is calculated by summing points and ranges from 0 to 14, with higher score representing higher adherence.
Change in the score for depression assessed by Zigmond and Snaith questionnaire to rate anxiety and depression | Baseline and at study completion at an average of 18 months, plus at the end of training (at an average of 12 to 15 months) in the intervention group
  Score achieved in the depression subscale of the Zigmond and Snaith test for anxiety or depression, a self-applied questionnaire. Depression scale includes 7 items each, scored on Likert scale from 0 to 3. Global score ranges from 0 to 21, with higher scores representing greater depression. The authors suggest that scores higher than eleven would indicate "case" and more than eight would be considered "probable case" (Zigmond and Snaith, 1983).
Change in the score for anxiety assessed by the Zigmond and Snaith questionnaire to rate depression and anxiety | Baseline and at study completion, plus at the end of training (at an average of 12 to 15 months) in the intervention group
  Score achieved in the anxiety subscale of the Zigmond and Snaith test for anxiety or depression, a self-applied questionnaire. Anxiety scale includes 7 items each, scored on Likert scale from 0 to 3. Global score ranges from 0 to 21, with higher scores representing greater anxiety. The authors suggest that scores higher than eleven would indicate "case" and more than eight would be considered "probable case" (Zigmond and Snaith, 1983).
Change in physical activity (minutes of dedicated physical activity) | Baseline and at study completion at an average of 18 months
  Minutes of In- and out-of-hospital dedicated physical activity
Change in physical activity assessed by the score in the Godin Leisure Test Exercise Questionnaire (GLTEQ) | Baseline and at study completion at an average of 18 months
  Score achieved in the Godin Leisure Test Exercise Questionnaire (GLTEQ) for quantification of physical activity. Activities are classified into three subgroups: "strenuous," "moderate," and "light." The scores corresponding to the energy expenditure (metabolic equivalent (MET)) are obtained by multiplying activities performed for more than 15 min in a week with their coefficients. The numbers represent the MET intensity values (strenuous/ exhausting exercises: 9 METs, moderate exercises: 5 METs, and light exercises: 3 METs).The increasing scores are associated with the increasing number of exercise behaviors, providing references about the contribution of physical activity to health: the activity score of 24 units and more as active (substantial benefits); the activity score of 14-23 units as moderately active (some benefits); and the activity score of 13 units and less as inactive (less substantial or low benefits).
Change in lymphedema assessed by perimeter of the upper limb by cirtometry (cm), stage and grade | Baseline after surgery and 2-4 weeks after the end of chemotherapy (at an average of 12 to 15 months)
  Perimeter of the upper limb by cirtometry (cm), stage and grade as defined by the Spanish Society of Rehabilitation and Physical Medicine

OTHER OUTCOMES:
Adherence and compliance to cardiac rehabilitation program (intervention group) assessed by number of training sessions attended/ number of sessions planned | At the end of the cardiac rehabilitation program at an average of 12 to 15 months
  Number of training sessions attended / number of sessions planned
Security of the cardiac rehabilitation program assessed by number of adverse events during training (intervention group) | At the end of the cardiac rehabilitation program at an average of 12 to 15 months
  Adverse events during training
Changes in expectations regarding the cardiac rehabilitation program assessed by a questionnaire (intervention group) | Baseline and at the end of the cardiac rehabilitation program at an average of 12 to 15 months
  Program-related expectations at baseline and at the end of the program' are collected through an open question "What do you expect to achieve by participating in the program?" Responses regarding expectations will be categorized by the evaluator within the following areas: psychological sphere and/or social sphere and/or physical sphere. Global expectations of benefit are scored from 0 (no benefit) to 10 (highest benefit).
Satisfaction with the cardiac rehabilitation program assessed by a questionnaire (intervention group) | At the end of the cardiac rehabilitation program at an average of 12 to 15 months
  Satisfaction at the end of the program is assessed by a questionnaire including 9 questions concerning comfort with training sessions, training spaces and development of the program, which are scored from 0 (worse posible result) to 10 (best posible result). Total score is calculated by adding for each question, and ranges from 0 to 90.
  * Due to the introduction of telematic exercise training during COVID-19 pandemic, questions were slightly modified to include assessment of satisfaction with this training modality.

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Martínez Monzonís, MD, PhD, Principal Investigator — Cardiology Department, Hospital Clínico Universitario de Santiago, CIBER-CV; Carlos Peña Gil, MD, PhD, Principal Investigator — Cardiology Department, Hospital Clínico Universitario de Santiago, CIBER-CV; José Ramón González Juanatey, MD, PhD, Study Director — Cardiology Department, Hospital Clínico Universitario de Santiago, CIBER-CV
Locations (1):
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain

REFERENCES:
- [Derived] Diaz-Balboa E, Gonzalez-Salvado V, Rodriguez-Romero B, Martinez-Monzonis A, Pedreira-Perez M, Cuesta-Vargas AI, Lopez-Lopez R, Gonzalez-Juanatey JR, Pena-Gil C. Thirty-second sit-to-stand test as an alternative for estimating peak oxygen uptake and 6-min walking distance in women with breast cancer: a cross-sectional study. Support Care Cancer. 2022 Oct;30(10):8251-8260. doi: 10.1007/s00520-022-07268-z. Epub 2022 Jul 11. PMID 35819522
- [Derived] Diaz-Balboa E, Gonzalez-Salvado V, Rodriguez-Romero B, Martinez-Monzonis A, Pedreira-Perez M, Palacios-Ozores P, Lopez-Lopez R, Pena-Gil C, Gonzalez-Juanatey JR. A randomized trial to evaluate the impact of exercise-based cardiac rehabilitation for the prevention of chemotherapy-induced cardiotoxicity in patients with breast cancer: ONCORE study protocol. BMC Cardiovasc Disord. 2021 Apr 7;21(1):165. doi: 10.1186/s12872-021-01970-2. PMID 33827450